CLINICAL TRIAL: NCT03797079
Title: Erector Spinae Plane Block Versus Thoracic Epidural Block as Analgesic Techniques for Chest Trauma
Brief Title: Erector Spinae Plane Block Versus Thoracic Epidural Block for Chest Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Fathy (Other)
Responsible Party: Sponsor-Investigator, Sameh Fathy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESP Block for Chest Trauma
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Chest Trauma
Keywords: Erector spinae plane block
MeSH Terms: conditions — Thoracic Injuries | interventions — Tea; Catheterization; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: The study subjects and the resident assessing the outcomes will be blinded to the study group. A single investigator will assess the patients for eligibility, obtain written informed consent, open the sealed opaque envelopes containing group allocation, perform the block, and administer bupivacaine solution.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (ESP block) (Active Comparator): Ultrasound-guided ESP block will be performed under strict aseptic precautions with patient in the sitting position. Catheter insertion will be performed and bupivacaine will be administered.
  Interventions: Procedure: ESP block; Device: Catheter insertion; Drug: Bupivacaine
- Group B (TEA) (Active Comparator): TEA will be performed under strict aseptic precautions with patient in the sitting position. Catheter insertion will be performed and bupivacaine will be administered.
  Interventions: Procedure: TEA; Device: Catheter insertion; Drug: Bupivacaine

INTERVENTIONS:
Procedure: ESP block — A high-frequency linear ultrasound probe will be placed superficial to erector spinae muscle (ESM) in a parasagittal plane 3 cm lateral to the midline at the level of fifth thoracic vertebra. Three muscles will be identified superficial to the hyperechoic transverse process shadow: trapezius (uppermost), rhomboids major (middle), and ESM (lowermost). After local infiltration of skin and using in-plane approach, an 18 G Tuohy needle will be inserted, until the tip lay between the rhomboid major muscle and ESM.
  Arms: Group A (ESP block)
Procedure: TEA — Skin will be locally infiltrated at the site of needle insertion, and 18 G Tuohy needle will be introduced until its tip lay in the epidural space of the T5-T6 thoracic intervertebral space.
  Arms: Group B (TEA)
Device: Catheter insertion — After obtaining loss of resistance, 20 G epidural catheter will be threaded for 5 cm and then fixed on the skin.
Drug: Bupivacaine — After the negative aspiration for blood, a bolus dose of 15 ml 0.125% plain bupivacaine will be injected in the catheter, followed by a continuous infusion of 0.25% plain bupivacaine at the rate of 0.1 ml/kg/h for 48 hours
  Other Names: Marcaine

SUMMARY:
Rib fractures are very common as a consequence of blunt chest trauma which is associated with severe pain, morbidity and mortality. The key to managing these patients is prompt and effective analgesia, early mobilization, respiratory support, with chest physiotherapy. The aim of this study is to compare and evaluate the differences between either continuous erector spinae plane (ESP) block, or thoracic epidural analgesia (TEA) as analgesic modalities in patients with chest trauma. It is hypothesized that ESP block will be comparable to TEA as a promising effective analgesic alternative with fewer side effects.

DETAILED DESCRIPTION:
Trauma is a major cause of morbidity and mortality worldwide as a leading cause of death. Rib fractures are very common and are detected in at least 10% of all injured patients, the majority of which are as a consequence of blunt chest trauma. Chest trauma are associated with severe pain, morbidity and mortality, as it contributes to atelectasis, lobar collapse, pneumonia, effusion, aspiration, acute respiratory distress syndrome pulmonary embolism, increased intensive care admissions, and poor overall clinical outcomes. Trauma is associated with release of cytokines, which contribute to the development of hemodynamic instability and metabolic derangement, which can worsen prognosis. The efficacy of utilizing different modalities for analgesia in controlling extent of tissue damage can be compared by measuring these cytokines levels. Multiple analgesic modalities have been used in these patients with chest trauma, such as oral analgesics, intravenous opioids, patient-controlled opioid analgesia, inter-pleural blocks, intercostal blocks, serratus plane blocks, paravertebral blocks, and TEA. In trauma patients with rib fractures, retrospective studies showed that TEA has become the gold standard of care, while ultrasound-guided paravertebral and serratus plane blocks are possible alternatives. However, no single best analgesic modality could be recommended or established, based on available data in this population, as no meta-analysis on this topic has yet been completed. Ultrasound has been the fundamental tool for a significant improvement in the progress of regional analgesic techniques of inter-fascial chest wall blocks, allowing their description and introduction into clinical practice. Ultrasound-guided ESP block is a new technique that has been recently described in the control of both chronic neuropathic pain as well as acute postsurgical or post-traumatic pain of the chest wall. The ESP block holds promise as a simple, easy, fast and safe technique for thoracic analgesia in the context of pain associated with chest trauma.

Aim of the Study:

The aim of this study is to assess the quality of pain relief and improvement of pulmonary function in patients with chest trauma receiving either continuous ESP block or TEA by comparing and evaluating the differences between the two techniques. It is hypothesized that ESP block will be comparable to TEA as a promising effective analgesic alternative with fewer side effects.

Sample Size Calculation:

The literature available on ESP block is limited to some sporadic case reports and editorials. Hence, this clinical trial will be conducted on 50 patients and post hoc analysis will be performed using pain scores obtained from the present study with an α (type I error) = 0.05 and β (type II error) = 0.2 (power = 80%).

Methods:

The study will be conducted in Mansoura Emergency Hospital on fifty patients admitted with chest trauma. They will be randomly assigned to two equal groups (ESP group and TEA group) according to computer-generated table of random numbers using the permuted block randomization method. The group allocation will be concealed in sequentially numbered, sealed opaque envelopes which will be opened only after obtaining the written informed consent. Patient demographic data including age, sex, body weight, and status of American Society of Anesthesiologists (ASA) will be recorded. A written informed consent will be obtained from all study subjects after ensuring confidentiality. The study protocol will be explained to all patients after enrollment into the study. In both groups, catheter-based analgesia will be performed with a bolus dose of bupivacaine followed by a continuous infusion for 48 hours. Later on, the catheters will be removed, and the pain management will be switched to parental or oral analgesics.

Statistical Methods:

The collected data will be coded, processed, and analyzed using Statistical Package for the Social Sciences (SPSS) program (version 22) for Windows. Normality of numerical data distribution will be tested by Shapiro-Wilk test. Continuous data of normal distribution will be presented as mean ± standard deviation, and compared with the unpaired student's t test. Non-normally distributed data will be presented as median (range), and compared with the Mann-Whitney U test. Repeated measures analysis of variance (ANOVA) test will be used for comparisons within the same group. Categorical data will be presented as number (percentage), and compared with the Chi-square test. All data will be considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) status: 1 or 2 .
* Blunt chest trauma.
* Multiple rib fractures.
* Flail chest.
* Lung contusions.

Exclusion Criteria:

* Bilateral chest trauma.
* Intubated patients.
* Other peripheral or abdominal injuries.
* Traumatic brain injury, altered mental status or un-cooperative patients.
* Acute spine fractures or pre-existing spine deformity.
* Unstable hemodynamics.
* Sensitivity to local anesthetic drugs.
* Coagulation abnormalities.
* Infection at the site of procedure.
* Significant cardiac or respiratory dysfunction, hepatic or renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Improvement in pain scores by Visual analogue scale (VAS) | Up to 48 hours after the procedure
  VAS score from 0 to 10 (0 = no pain and 10 = the worst imaginable pain) will be assessed every two hours for 48 hours after the procedure.

SECONDARY OUTCOMES:
Total analgesic requirements of fentanyl | Up to 48 hours after the procedure
  The amount of fentanyl consumption given as a rescue analgesia to patients will be measured all over the 48 hours.
First analgesic request | Up to 48 hours after the procedure
  The time of the first analgesic request for fentanyl will be recorded.
Changes in heart rate (HR) | Up to 48 hours after the procedure
  HR will be recorded every two hours for 48 hours after the procedure.
Changes in mean arterial blood pressure (MAP) | Up to 48 hours after the procedure
  MAP will be recorded every two hours for 48 hours after the procedure.
Improvement in forced expiratory volume in one second (FEV1) | Up to 48 hours after the procedure
  FEV1 will be assessed by spirometry before and 48 hours after the procedure.
Improvement in forced vital capacity (FVC) | Up to 48 hours after the procedure
  FVC will be assessed by spirometry before and 48 hours after the procedure.
Improvement in forced expiratory flow (FEF 25-75%) | Up to 48 hours after the procedure
  FEF 25-75% will be assessed by spirometry before and 48 hours after the procedure.
Improvement in the level of tumor necrosis factor alpha (TNF-α) | Up to 48 hours after the procedure
  TNF-α will be measured before, 24, 48 hours after the procedure.
Improvement in the level of interleukin 6 (IL-6) | Up to 48 hours after the procedure
  IL-6 will be measured before, 24, 48 hours after the procedure.
Incidence of adverse effects | Up to 48 hours after the procedure
  Any adverse effects like pneumothorax, respiratory depression, nausea, vomiting, hematoma, or allergic reactions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M El-Sherbiny, MD, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Gage A, Rivara F, Wang J, Jurkovich GJ, Arbabi S. The effect of epidural placement in patients after blunt thoracic trauma. J Trauma Acute Care Surg. 2014 Jan;76(1):39-45; discussion 45-6. doi: 10.1097/TA.0b013e3182ab1b08. PMID 24368355
- [Background] Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, Shaefer G, To KB, Fox AD, Alley DE, Ditillo M, Joseph BA, Robinson BR, Haut ER. Pain management for blunt thoracic trauma: A joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. J Trauma Acute Care Surg. 2016 Nov;81(5):936-951. doi: 10.1097/TA.0000000000001209. PMID 27533913
- [Background] Nagaraja PS, Ragavendran S, Singh NG, Asai O, Bhavya G, Manjunath N, Rajesh K. Comparison of continuous thoracic epidural analgesia with bilateral erector spinae plane block for perioperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):323-327. doi: 10.4103/aca.ACA_16_18. PMID 30052229
- [Background] Singh S, Jacob M, Hasnain S, Krishnakumar M. Comparison between continuous thoracic epidural block and continuous thoracic paravertebral block in the management of thoracic trauma. Med J Armed Forces India. 2017 Apr;73(2):146-151. doi: 10.1016/j.mjafi.2016.11.005. Epub 2016 Dec 24. PMID 28924315
- [Background] Veiga M, Costa D, Brazao I. Erector spinae plane block for radical mastectomy: A new indication? Rev Esp Anestesiol Reanim (Engl Ed). 2018 Feb;65(2):112-115. doi: 10.1016/j.redar.2017.08.004. Epub 2017 Nov 2. English, Spanish. PMID 29102405
- [Background] Witt CE, Bulger EM. Comprehensive approach to the management of the patient with multiple rib fractures: a review and introduction of a bundled rib fracture management protocol. Trauma Surg Acute Care Open. 2017 Jan 5;2(1):e000064. doi: 10.1136/tsaco-2016-000064. eCollection 2017. PMID 29766081
- [Background] Yeh DD, Kutcher ME, Knudson MM, Tang JF. Epidural analgesia for blunt thoracic injury--which patients benefit most? Injury. 2012 Oct;43(10):1667-71. doi: 10.1016/j.injury.2012.05.022. Epub 2012 Jun 16. PMID 22704784